CLINICAL TRIAL: NCT06778148
Title: Abridge AI Pilot Test
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 24-1623
Record Dates: First submitted 2025-01-10; First posted 2025-01-16 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Clinician Experience; Clinician Burnout
Keywords: Ambient AI; Clinician burnout

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with waitlist
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Assigned Abridge license (Experimental): Providers assigned a license
  Interventions: Other: Ambient AI for clinician documentation
- Control (No Intervention): Providers not assigned a license or waitlisted

INTERVENTIONS:
Other: Ambient AI for clinician documentation — Ambient AI for clinician documentation
  Other Names: Abridge
  Arms: Assigned Abridge license

SUMMARY:
We are piloting a new technology (Abridge) that uses artificial intelligence to listen to clinician-patient office visits and then document the interaction in the electronic health record.

DETAILED DESCRIPTION:
This study will evaluate pilot implementation of the Abridge Artificial Intelligence (AI) Platform (Abridge) in UCHealth clinics. Abridge licenses will be deployed to 116 physician and advanced practice clinicians to accomplish the following goals:

1. Determine if Abridge meaningfully impacts clinician documentation time and burnout or stress
2. Determine whether to scale Abridge beyond the pilot

We will evaluate clinician experiences using Abridge, particularly with regard to documentation time and clinician burnout or stress. Study findings will explore value added in integrating Abridge into clinician practice, and guide decision-making for entering into a commercial agreement with Abridge. This pilot will also inform best practices for scaling Abridge to a broader user base across UCHealth outpatient practices.

ELIGIBILITY:
Inclusion Criteria:

-clinician (physician, advance practice professional, or licensed mental health professional) employed by UCHealth

* See clinic patients at least three half-day sessions per week. (Half-day sessions seeing or supervising patients with residents and fellows will NOT count toward the weekly total. Half-day sessions seeing patients with a medical student CAN count toward the weekly total, however, Abridge can only capture conversations where you are physically present with patients.)
* Own an iOS smartphone and be willing to download and use the Epic Haiku smartphone app during clinic visits

Exclusion Criteria:

* Trainees including residents and fellows
* PT/OT, ED, maternal/fetal, pediatric, dental, eye specialties

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2025-07-13 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Burnout - High emotional exhaustion | Baseline, 2, 4 and 8 months
  Validated measure collected by survey. Reference: https://pmc.ncbi.nlm.nih.gov/articles/PMC3475833/
Burnout - High depersonalization | Baseline, 2, 4 and 8 months
  Validated measure collected by survey. Reference: https://pmc.ncbi.nlm.nih.gov/articles/PMC3475833/
Burnout - emotional exhaustion and depersonalization | Baseline, 2, 4 and 8 months
  Validated measure collected by survey. Reference: https://pmc.ncbi.nlm.nih.gov/articles/PMC3475833/
Time in notes per appointment | Baseline, 2, 4 and 8 months
  Collected via EHR signal data
Adoption | 2, 4 and 8 months
  Percent of eligible visits in which intervention is used. Collected via EHR data

SECONDARY OUTCOMES:
Reach | 2, 4 and 8 months
  Proportion and representativeness of eligible patients and visits intervention was used for
Clinician experience | Baseline, 2, 4 and 8 months
  Likelihood to recommend via validated NPS, qualitative drivers of experience, likelihood to change jobs, Weiners feasiblity/implementability/acceptability, system usability scale
Time documenting | Baseline, 2, 4 and 8 months
  Time spent documenting beyond appointment, average time in the EHR, time of last log out of the day, pajama time documenting
Operational efficiency | Baseline, 2, 4 and 8 months
  Same day note closure, average note star rating, average note turn around time
Adoption | 2, 4 and 8 months
  Abandonment rate and representativeness

CONTACTS AND LOCATIONS:
Locations (1):
- UCHealth, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
Unsure if the third party owner of Abridge will allow sharing